CLINICAL TRIAL: NCT00207649
Title: Shared Decision Making: Prostate Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Richarson (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Lisa Richarson, Associate Director for Science, Centers for Disease Control and Prevention
Organization: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: CDC-NCCDPHP-R-01-PH-000019
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: shared decision-making; prostate cancer screening; evidence-based medicine; computer-assisted learning tools; standardized patients; randomized controlled trial; educational intervention; patient education; physician education
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): standard informational brochures
- Web curriculum for physicians only (Experimental): Both intervention arms will use a novel web-based interactive curriculum that provides education about prostate cancer screening, including potential benefits and harms, fundamentals of effective patient counsel, and shared decision-making. In one of the intervention arms, the physicians saw the web-based interactive curriculum and the patient received the brochure.
  Interventions: Behavioral: Shared decision-making for PSA screening tool
- Web curriculum for physicians and patients (Experimental): In the other intervention arm, the physicians saw the web-based curriculum and the patient received interactive curriculum covering content similar to that contained in the web-based interactive curriculum for physicians.
  Interventions: Behavioral: Shared decision-making for PSA screening tool

INTERVENTIONS:
Behavioral: Shared decision-making for PSA screening tool — Interventions to Improve Shared Decision-Making: Prostate Cancer Screening is a prospective study of educational interventions to improve shared decision-making of physicians and their patients about prostate cancer screening. Physicians will be randomized by practice site to receive standard informational brochures (control group) or a novel web-based interactive curriculum that provides education about prostate cancer screening, including potential benefits and harms, fundamentals of effective patient counsel, and shared decision-making. In addition, patients at intervention sites will be randomized to receive either the brochure or a patient-oriented interactive curriculum covering content similar to that contained in the physician tool. Physicians in all groups will also see one unannounced standardized patient (SP) trained to portray a patient interested in discussing PSA.
  Arms: Web curriculum for physicians and patients; Web curriculum for physicians only

SUMMARY:
Interventions to Improve Shared Decision-Making: Prostate Cancer Screening is a prospective study of educational interventions to improve the interaction of physicians and their patients about prostate cancer screening. Educational material is provided in primary care practices using either standard paper information or a novel web-based interactive curriculum that explores the risks and benefits of screening measures for prostate cancer for older men. The impact of the intervention on shared decision-making with both actual and standardized patients will be assessed.

DETAILED DESCRIPTION:
Prostate cancer is an important cause of death and disability in US men, but the value of screening for the disease with the prostate specific antigen (PSA) test remains highly controversial. Many primary care physicians use PSA testing routinely, with little patient counseling. Interventions to Improve Shared Decision-Making: Prostate Cancer Screening is a prospective study of educational interventions to improve shared decision-making of physicians and their patients about prostate cancer screening. Physicians will be randomized by practice site to receive standard informational brochures (control group) or a novel web-based interactive curriculum that provides education about prostate cancer screening, including potential benefits and harms, fundamentals of effective patient counsel, and shared decision-making. In addition, patients at intervention sites will be randomized to receive either the brochure or a patient-oriented interactive curriculum covering content similar to that contained in the physician tool. The intervention will be evaluated among 140 physicians within a variety of primary care settings (i.e., University-based clinics, staff-model managed care clinics, and military affiliated outpatient clinics). Approximately 10-15 actual patients of each participating physician will complete a post-visit questionnaire describing their discussion with their doctor about prostate cancer, PSA, and their decision about whether to be screened. Physicians in all groups will also see one unannounced standardized patient (SP) trained to portray a patient interested in discussing PSA. Study groups will be compared on the extent of shared decision-making they engage in with both actual and standardized patients. Pre- and post-study changes in physician knowledge and attitudes about PSA as well as the physicians' pre- and post-study PSA test ordering rates will be ascertained.

ELIGIBILITY:
Inclusion Criteria:

* Physicians in primary care practice settings with male patients age 50-75

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Intervention groups (physician education only, both physician and patient education) vs. control group comparison of physician shared decision-making (SDM) behaviors (self-reported SDM and SDM reported by actual and standardized patients) | study period

SECONDARY OUTCOMES:
1.Pre- and post-study changes in physician knowledge and attitudes about PSA | study period
2.Pre- and post-study changes in physicians' PSA ordering behavior for their patients age 50-75 years | study period
3.Patients post-visit knowledge and attitudes about PSA | study period

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Wilkes, MD PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Center for Health Services Research, Sacramento, California, United States